CLINICAL TRIAL: NCT07148973
Title: Outcomes for Patients With Ascending Aortic Dilation Who Underwent Transcatheter Aortic Valve Replacement in a Chinese Population
Brief Title: Outcomes for Patients With Ascending Aortic Dilation Who Underwent TAVR
Status: Completed | Type: Observational
Sponsor: zjq (Other)
Responsible Party: Sponsor-Investigator, zjq, Investigator, Affiliated Zhongshan Hospital of Dalian University
Organization: Affiliated Zhongshan Hospital of Dalian University (Other)
Other Study IDs: 2021062
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Transcatheter Aortic Valve Replacement (TAVR); Ascending Aortic Dilation
MeSH Terms: conditions — Aneurysm, Ascending Aorta | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- AAD
  Interventions: Procedure: Transcatheter Aortic Valve Replacement

INTERVENTIONS:
Procedure: Transcatheter Aortic Valve Replacement — The TAVR surgery mainly involves attaching an artificially-made aortic valve to a special catheter, and then using the catheter to deliver the valve to the affected area and release it. This surgery replaces the original aortic valve with an artificial one, thereby restoring the valve function. Compared with traditional open-chest surgery, it causes less trauma, has lower risks, and enables faster recovery. It is particularly suitable for patients who cannot tolerate open-chest surgery, have poor cardiac function, or are older.

SUMMARY:
The present study was designed to evaluate the safety of TAVR with a preoperative ascending aortic (AA) diameter ≥ 40 mm. This study also aimed to explore the procedural outcomes and clinical prognoses of patients with AAD combined compared to those of patients without AAD combined who underwent TAVR.

Between January 2019 and July 2021, a total of 186 patients who were diagnosed at a single centre with severe AS underwent the TAVR procedure using a self-expanding valve. The AA diameter was evaluated via 3-dimensional (3D) multidetector computed tomography (MDCT) before TAVR. AAD was defined as a value of AAD ≥ 40 mm.

ELIGIBILITY:
Inclusion Criteria:

* (1) severe AS patients diagnosed on the recommendation of the European Society of Cardiology/European Association for Cardio-Thoracic Surgery Guidelines (aortic valve area ≤ 1.0 cm²/aortic valve index ≤ 0.6 cm²/m²/peak aortic velocity (Vmax)≥4.0 m/s); (2) patients at intermediate- to high-risk surgical risk or a Society of Thoracic Surgeons risk (STS) score > 4; (4) patients whose anatomy was evaluated by 3-dimensional (3D) multidetector computed tomography (MDCT) appropriate for TAVR; and (4) patients with severe AS with typical symptoms.

Exclusion Criteria:

* (1) patients with active endocarditis, acute aortic dissection, or acute myocardial infarction; (2) patients with expectations of life< 1 year; and (3) patients with inappropriate anatomy evaluated by 3D MDCT.

Ages: 50 Years to 93 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who were diagnosed with severe AS via the TAVR procedure using a self-expanding valve (Venus-A valve, Qiming Med Tech Inc., Hangzhou, China) between January 2019 and July 2021 at our Heart Center were retrospectively enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

PRIMARY OUTCOMES:
All-Cause Mortality | 6 month
Mortality | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- the Affiliated Zhongshan Hospital of Dalian University, Dalian, Liaoning, China

IPD SHARING:
Plan to Share IPD: Undecided